CLINICAL TRIAL: NCT05031390
Title: the Horsens Aarhus FemoroAcetabular Impingement Syndrome Training Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horsens Hospital (Other)
Collaborators: University of Aarhus (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, Jeppe Lange, Head of Research, Horsens Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-16-02-724-18
Record Dates: First submitted 2021-08-12; First posted 2021-09-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapist-led training (Experimental): Physiotherapy-led training of patients with FAIS
  Interventions: Procedure: Physiotherapist-led training

INTERVENTIONS:
Procedure: Physiotherapist-led training — Patients will undergo a 12-week physiotherapist-led training program consisting of 8 supervised sessions and home-based training in between

SUMMARY:
The aim of the study is to investigate the feasibility of a training intervention in patients with femoroacetabular impingement syndrome (FAIS).

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility of a 12-weeks (progressive) exercise program in patients with FAIS. Feasibility is evaluated on the recruitment strategy, patient adherence to the exercises and their experiences with and motivation for performing exercises. Furthermore, the investigators wish to investigate the variation of data before and after the exercise program to help estimate a suitable sample size for a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-50 years old
2. Diagnosed with FAIS according to the Warwick agreement
3. Patients having cam morphology should have an alpha angle of > 55 degrees on an anterior-posterior radiograph.
4. Patients having pincer should have a lateral centre edge angle of >39 degrees on an anterior-posterior radiograph.
5. Lateral joint space width should be >3 mm.
6. Body mass index is below 30.
7. Motivated for participation in a 12 week training program with 8 physical attendances.

Exclusion Criteria:

1. Received physiotherapist-led treatment in the past 3 months,
2. Previous hip surgery in included hip or other major hip injury,
3. Systemic conditions e.g. rheumatoid arthritis, cancer,
4. Chronical pain syndromes,
5. Unable to perform testing procedures,
6. Unable to attend a 12-week treatment program or baseline and follow-up assessments
7. Contraindications to radiographs (e.g. pregnancy)
8. Unable to read or understand questionnaires and/or instructions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Number of completed exercise sessions | 0-12 weeks
  Number of completed exercise sessions. A high adherence is defined as attendance of > 75% of planned sessions
Completion of training program | 0-12 weeks
  The training program is considered completed if patients are not dropping out of the study before the end of the 12 weeks. Completion rate will be calculated as % patients who completed the study

SECONDARY OUTCOMES:
The Copenhagen Hip and Groin Outcome Score (HAGOS) | Change from 0-12 weeks
  HAGOS is a questionnaire developed for young, active persons experiencing hip and/or groin pain. It consists of 6 subscales: Pain, Symptoms, Activities of Daily Living, Sport, Participation in Sport and Hip-related quality of life. The main subscales used in this study are HAGOS pain and sport.
The International Hip Outcome Tool (iHOT-33) | Change from 0-12 weeks
  iHOT-33 is a questionnaire focussing at patients' hip related quality of life in 33 questions. Both a total score and sub scales: "Symptoms and functional limitations", "Sports and recreational activities", "Job related concerns" and "Social, emotional and lifestyle concerns", are extracted from the questionnaire.
The Hip Sports Activity Scale (HSAS) | Change from 0-12 weeks
  Current physical activity measured from 0 to 8 points, 0 being no activity and 8 being an athlete
Maximal hip muscle strength | Change from 0-12 weeks
  Change (Nm/kg) in maximal hip flexion, extension, abduction and adduction from 0-12 weeks
One-legged hop for distance | 0-12 weeks
  Change (cm) i hop distance from 0-12 weeks
Y-balance board | 0-12 weeks
  Change (cm) in ability to perform on the y balance board from 0-12 weeks
Patient Acceptable Symptom State | 0-12 weeks
  Patient Acceptable Symptom State (yes/no): Change in number of patients reporting yes vs. no from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Signe Kierkegaard, PhD, Principal Investigator — Regionshospitalet Horsens
Locations (1):
- Signe Kierkegaard, Horsens, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Pilot study with few participants.